CLINICAL TRIAL: NCT01083160
Title: Clinical Outcomes,Compliance and Effectiveness of Switching From Infliximab or Etanercept to Adalimumab. A Multicenter Post-Marketing Observational Study in Routine Clinical Use
Brief Title: Clinical Outcomes, Compliance and Effectiveness of Switching From Infliximab or Etanercept to Adalimumab in Patients With Active Rheumatoid Arthritis (RA). A Multicenter Post-Marketing Observational Study in Routine Clinical Use
Acronym: FALLA
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to low enrollment because inclusion criteria are obsolete.
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-604
Record Dates: First submitted 2010-02-19; First posted 2010-03-09 (Estimated); Results first posted 2012-01-02 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anti-TNF; Adalimumab; Infliximab; Etanercept
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Non responders to other anti-TNF: Patients with lack of efficacy to infliximab or etanercept treated with adalimumab according to the routine clinical practice of the participating centers. A 40 mg dose was administered every other week for 24 weeks.

SUMMARY:
This is a prospective, single-arm, post marketing observational study in adult patients with active rheumatoid arthritis (RA) who are discontinuing treatment due to lack of efficacy, intolerance or to an incomplete response with either infliximab or etanercept.

The aim of this post-marketing observational study is to obtain data on clinical outcomes, compliance and tolerability to determine the effectiveness of switching from infliximab or etanercept to adalimumab. In this cohort, the different treatment strategies are to be studied in the context of the routine clinical practice in the different participating places.

DETAILED DESCRIPTION:
This is a prospective, single-arm, post marketing observational study in adult patients with active RA who are discontinuing treatment due to lack of efficacy, intolerance or to an incomplete response with either infliximab or etanercept.

The aim of this post-marketing observational study is to obtain data on clinical outcomes, compliance and tolerability to determine the effectiveness of switching from infliximab or etanercept to Adalimumab. In this cohort, the different treatment strategies are to be studied in the context of the routine clinical practice in the different participating places.

Study Objectives:

Primary objective:

To assess the effectiveness of the treatment with adalimumab in patients with rheumatoid arthritis (RA) that have failed or presented an incomplete response to current treatment with either infliximab or etanercept.

Secondary objective:

To evaluate the compliance and clinical tolerability with adalimumab

Investigational Plan and Selection of Study Population:

All patients belonging to any of the centres participating in the study that meet all the inclusion criteria and none of the exclusion criteria will be considered eligible.

Patients considered eligible for the study will have to give their consent for the use and/or disclose of the patient's personal and/or health data. Patient's consent will be obtained before his/her participation in the study and will be documented in an Informed Consent Form approved by an Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 and <75 years of age that meet the American College of Rheumatology (ACR) criteria for RA.
* Patients with active RA defined as:

  1. ≥3 tender joints and ≥3 swollen joints, or
  2. DAS 28 score >3.1
* Patients who are discontinuing treatment with either infliximab or etanercept due to:

  1. Lack of efficacy, or
  2. Incomplete response.
* Patients that, in the opinion of the physician could result beneficiated with the locally approved treatment scheme of adalimumab
* Those patients who switch from infliximab or etanercept to adalimumab has been done in the last 60 days could be included in the study.

Exclusion Criteria:

The following patients will not be included in the study:

* Patients who have active infections.
* Patients with latent TB. For this protocol, evidence of latent TB infection is defined as an induration (not erythema) of 5 mm or greater, 48-72 hrs after placement. Any suggested data on the clinical history or chest x-ray.
* Patients participating into another study or clinical trial
* Any condition that according to the criteria of the participating physician represents an obstacle for study conduct and/or represents a potential unacceptable risk for patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2008-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pozos, MD, Study Chair — Abbott
Locations (12):
- Mexico (12):
  - Site Reference ID/Investigator# 27882, Chihuahua City
  - Site Reference ID/Investigator# 27883, Chihuahua City
  - Site Reference ID/Investigator# 27884, Culiacán Sin.
  - Site Reference ID/Investigator# 27888, Guadalajara, Jal.
  - Site Reference ID/Investigator# 27886, Guadalajara, Jal.
  - Site Reference ID/Investigator# 27887, Guadalajara, Jal.
  - Site Reference ID/Investigator# 25943, Leon, Gto.
  - Site Reference ID/Investigator# 28059, Mexico City
  - Site Reference ID/Investigator# 27885, Mexico City
  - Site Reference ID/Investigator# 27890, Puebla, Pue.
  - Site Reference ID/Investigator# 27889, Puebla, Pue.
  - Site Reference ID/Investigator# 28057, Tuxtla Gutiérrez

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non Responders to Other Anti-TNF
Started | 82
Evaluable Population | 71
Completed | 81
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Non Responders to Other Anti-TNF
Number analyzed (Participants) | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 48.34 (11.56)
Sex/Gender, Customized [Number; unit: participants]
  Female | 66
  Male | 13
  Gender not reported | 3
Region of Enrollment [Number; unit: participants]
  Mexico | 82

OUTCOME MEASURES:

1. Primary Outcome: DAS28 (Disease Activity Score in 28 Joints)
Description: The DAS 28 index measures disease activity in rheumatoid arthritis and is derived from the number swollen/tender joints, laboratory tests of inflammation, and participant assessment of global health (by marking a 10 cm line from "very good" to "very bad"). Ranges were used to classify participants, with a higher score indicating worse control of disease: Remission (<= 2.6), Low Disease Activity (>2.6 to <=3.2), Moderate Disease Activity (>3.2 to <= 5.1) and High Disease Activity (>5.1). The mean change in DAS 28 score from baseline to each visit is presented.
Time Frame: Baseline and Weeks 8,16 and 24
Population: Analysis conducted in participants with results at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non Responders to Other Anti-TNF
Number analyzed (Participants) | 82
units on a scale
  DAS 28 at Baseline (n=82) | 6.04 (1.17)
  DAS 28 at Week 8 (n=80) | 4.63 (1.77)
  DAS 28 at Week 16 (n=79) | 4.05 (1.74)
  DAS 28 at Week 24 (n=71) | 3.68 (1.47)

2. Primary Outcome: Tender Joint Count and Swollen Joint Count
Description: The treating physician was to clinically assess each participant at each study visit and report the number of tender and swollen joints. The mean number of painful or swollen joints for participants evaluated at each time point are presented.
Time Frame: Baseline and Weeks 8,16 and 24
Population: Analysis conducted in participants with results at each time point.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Non Responders to Other Anti-TNF
Number analyzed (Participants) | 82
Joints
  Tender joints at Baseline (n=82) | 13.05 (7.29)
  > Week 8 (n=80) | 7.16 (6.37)
  >Week 16 (n=80) | 5.44 (5.76)
  >Week 24 (n=71) | 4.23 (5.32)
  Swollen joints at Baseline (n=82) | 9.56 (5.97)
  >Week 8 (n=80) | 4.48 (4.68)
  >Week 16 (n=80) | 3.15 (4.67)
  >Week 24 (n=71) | 2.52 (4.10)

3. Primary Outcome: Severity of Pain in a 100mm Visual Analogue Scale (VAS 100mm)
Description: Participants assessed the severity of their pain using a 0 to 100 mm horizontal visual analogue scale (VAS). The far left end indicated no pain (0 mm) and the far right meant the worst possible pain (100 mm). Participants drew a vertical line on the horizontal scale to indicate their current level of pain at each visit.
Time Frame: Baseline and Weeks 8,16 and 24
Population: Analysis conducted in participants with results at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Non Responders to Other Anti-TNF
Number analyzed (Participants) | 82
Units on a scale
  VAS at Baseline (n=82) | 62.88 (22.31)
  >Week 8 (n=80) | 39.69 (25.40)
  >Week 16 (n=80) | 32.35 (26.02)
  >Week 24 (n=71) | 28.70 (23.32)

4. Secondary Outcome: Evaluate the Compliance and Clinical Tolerability With Adalimumab
Description: To assess compliance, participants were asked at the Week 8 and Week 16 visits how many doses they had missed since their previous visit. Adverse events were collected throughout the study, from the time the participant signed the informed consent form until 30 days or 5 half-lives after the last dose of study drug. For additional information see the Reported Adverse Event section.
Time Frame: Baseline to Week 24
Population: Analysis population included all participants enrolled in the study who took at least one dose of adalimumab.
Measure: Number; unit: Participants
Arm/Group | Non Responders to Other Anti-TNF
Number analyzed (Participants) | 82
Participants
  Reported 1 missed dose at Week 8 | 1
  Reported 2 missed doses at Week 8 | 3
  Reported 2 missed doses at Week 16 | 1
  Reported 3 missed doses at Week 16 | 1
  Experienced a non-serious adverse event | 6
  Experienced a serious adverse event | 1

ADVERSE EVENTS:
Time Frame: Duration of study participation was 24 weeks. Adverse events were collected from the time the participant signed the informed consent form until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment.
Arm/Group | Non Responders to Other Anti-TNF
Serious Adverse Events (participants affected / at risk) | 1/82
Other Adverse Events (participants affected / at risk) | 6/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Responders to Other Anti-TNF (N=82)
rectal bleeding (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Responders to Other Anti-TNF (N=82)
Constipation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Phosphenes (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Swelling in administration site (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection